CLINICAL TRIAL: NCT06617312
Title: Examining the Effects of Cytisinicline on Neural Substrates of Cigarette Cue-Reactivity
Acronym: Cytisinicline
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Lara Ray, PhD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-001071; T34FT8089 (Other: Tobacco Related Disease Research Program)
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Smoking Cessation; Tobacco Use Disorder
Keywords: smoking cesstion; tobacco use disorder; cigarette smoking; fMRI; cytisinicline
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder; Cigarette Smoking | interventions — cytisine

STUDY DESIGN:
Intervention Model Description: We will randomize 64 non-treatment seeking adults who smoke cigarettes (N=32 cytisinicline, N=32 placebo; 50% females) in a double-blind, placebo-controlled laboratory study testing the effects of cytisinicline on the neural substrates of cigarette cue reactivity. All participants will be daily combustible cigarette smokers. Interested individuals will call the lab and complete a telephone screening interview. Individuals who are deemed eligible will receive a full explanation of study procedures and provide written, informed consent. Participants will then complete a behavioral screen and physical exam. Eligible participants will then be randomized to a medication, cytisinicline (3 mg, 3 times daily) or placebo (0mg, 3 times daily). Participants will complete brief daily diary self-reports of cigarette use and craving during the outpatient medication period. Following 2- to 3-weeks of cytisinicline, or placebo, treatment participants will complete a cigarette cue-exposure fMRI task.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cytisinicline (Experimental): 3mg cytisinicline oral capsule 3 times daily for 2-to-3 weeks
  Interventions: Drug: Cytisinicline
- Placebo (Placebo Comparator): matched to experimental drug
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Cytisinicline — Targets α4β2 nicotinic acetylcholine receptors
  Arms: Cytisinicline
Drug: Placebo Oral Capsule — Matched to active drug, cytisinicline
  Arms: Placebo

SUMMARY:
This study will randomize 64 non-treatment seeking individuals who smoke cigarettes daily in a double-blind, placebo-controlled laboratory study testing the effects of cytisinicline on the neural substrates of cigarette cue reactivity.

DETAILED DESCRIPTION:
The objective of this study is to examine the effects of cytisinicline on neural substrates of cigarette cue-reactivity. We will randomize 64 adults who smoke cigarettes daily (N=32 cytisinicline, N=32 placebo; 50% female) into a double-blind, placebo-controlled laboratory study of cytisinicline. Specifically, participants will complete a 2- to 3-week outpatient protocol that includes taking cytisinicline (3 mg, 3 times daily) or matched placebo (0 mg, 3 times daily) and completing a brief daily diary assessment of cigarette use and craving. Following 2- to 3-weeks of cytisinicline (or placebo) treatment, participants will complete a cigarette cue-exposure task during fMRI. Total study participation will be approximately 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. be between the ages of 18 and 65 and provide informed consent;
2. smoke 5 or more combustible cigarettes per day;
3. not seeking treatment for smoking;

Exclusion Criteria:

1. current use of other smoking cessation aid (bupropion, varenicline, nortriptyline, NRT);
2. more than 3 months of smoking abstinence in past year;
3. use of non-cigarette tobacco product (pipe tobacco, cigars, smokeless tobacco, hookah) or electronic cigarettes more than 5 times in the 28-days prior to enrollment;
4. current use of psychoactive drug (excluding cannabis), as determined by urine toxicology;
5. current (past 12-month) DSM-5 diagnosis of substance use disorder for any substances other than tobacco and mild cannabis or mild-to-moderate alcohol use disorders;
6. lifetime history of psychotic disorders, bipolar disorders, or major depression with suicidal ideation;
7. current suicidal ideation or lifetime history of suicide attempt;
8. serious medical illness within past 3 months, including recent history of acute myocardial infarction, unstable angina, stroke, cerebrovascular incident, or hospitalization for congestive heart failure;
9. medical condition that may interfere with safe study participation;
10. renal impairment defined as a creatinine clearance (CrCl) greater than 60 mL/min (estimated with the Cockroft-Gault equation);
11. exceed Grade 2 laboratory abnormalities, based on FDA Guidance Document "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials";
12. uncontrolled hypertension (blood pressure ≥160/100 mmHg);
13. abnormal electrocardiogram;
14. non-removable ferromagnetic object in body;
15. claustrophobia;
16. serious head injury or period of unconsciousness (more than 30 minutes);
17. more than 250lbs;
18. Be pregnant, nursing, or planning to become pregnant while taking part in the study; and must agree to one of the following methods of birth control (if female), unless she or partner are surgically sterile:

    * Oral contraceptives
    * Contraceptive sponge
    * Patch
    * Double barrier
    * Intrauterine contraceptive device
    * Etonogestrel implant
    * Medroxyprogesterone acetate contraceptive injection
    * Hormonal vaginal contraceptive ring
    * Complete abstinence from sexual intercourse;
19. have experienced adverse effects to varenicline;
20. have an intense fear of needles or have had an adverse reaction to needle puncture.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Blood-oxygen-level-dependent (BOLD) activation to cigarette cues during fMRI task | From enrollment to end of treatment at 2-to-3 weeks
  Participants will complete a cigarette cue-exposure task during fMRI. In this paradigm, participants are exposed to videotaped cues of smoking and control, non-cigarette related, content. Blood-oxygen-level-dependent (BOLD) activation to cigarette (vs. non-cigarette control ) cues will be calculated.

SECONDARY OUTCOMES:
In-scanner cigarette cue-induced subjective craving | From enrollment to end of treatment at 2-to-3 weeks
  In-scanner cigarette cue-induced subjective craving ratings will be obtained following each cue exposure during the fMRI task.
Subjective cigarette craving during outpatient period | From enrollment to end of treatment at 2-to-3 weeks
  Subjective cigarette craving, as assessed via daily diary self-report assessments, during the outpatient medication period

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States